CLINICAL TRIAL: NCT01339078
Title: Randomized Controlled Trial Comparing Kaffes Stent With Plastic Prosthesis in the Treatment of Anastomotic Biliary Strictures Post Orthotopic Liver Transplantation
Brief Title: Trial Comparing Kaffes Stent With Plastic Prosthesis in the Treatment of Anastomotic Biliary Strictures Post Orthotopic Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/255
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Biliary Strictures Post Liver Transplantation
Keywords: Biliary strictures; liver transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plastic stenting (Active Comparator): Patients will be randomized towards plastic stenting.
  Interventions: Procedure: Plastic stenting
- Kaffes stenting (Experimental): Patients will be randomized towards Kaffes stenting.
  Interventions: Procedure: Kaffes stenting

INTERVENTIONS:
Procedure: Plastic stenting — The patients receive plastic stenting after ortothopic liver transplantation with a choledocho-choledochal anastomosis, presenting with an anastomotic stricture. These patients will receive change of the stent every 3 months, for a total duration of 1 year.
  Arms: Plastic stenting
Procedure: Kaffes stenting — The patients receive Kaffes stenting after ortothopic liver transplantation with a choledocho-choledochal anastomosis, presenting with an anastomotic stricture. These patients will receive change of the stent every 6 months, for a total duration of 1 year.
  Arms: Kaffes stenting

SUMMARY:
Biliary anastomotic strictures (post liver transplantation) occur in 15-20 % of the cases. Biliary stenting using plastic prosthesis during a period of 1 year is the treatment of choice. Problematic in this approach is the regular change, necessary to overcome occlusion of the stent, resulting in cholestasis and/or infection. This change needs to be performed every 3 months or more frequently in patients with symptoms of stent occlusion.

The Kaffes stent (RMS) is a metallic removable stent, especially constructed for the treatment of biliary anastomotic strictures post liver transplantation. The advantage could be that this stent is less prone to occlusion with a lower change frequency (e.g. every 6 months).

No randomized, controlled trial (RCT) or data exist comparing plastic stenting versus Kaffes stenting.

ELIGIBILITY:
Inclusion Criteria:

* Patients after orthotopic liver transplantation with a choledocho- choledochal anastomosis, presenting with an anastomotic stricture
* diagnosis established by :

  * elevated liver tests
  * a narrowing of the anastomosis on Magnetic resonance cholangiopancreatography (MRCP): with or without intrahepatic bile duct dilatation
  * no acute or chronic rejection
  * no Cytomegalovirus (CMV) infection
  * no other possible causes of elevated liver tests
  * confirmation of the stricture needs to be confirmed during the diagnostic endoscopic retrograde cholangiopancreatography (ERCP) procedure immediately before the therapeutic procedure.

Exclusion Criteria:

* non-anastomotic strictures
* absence of informed consent
* Roux-en-Y construction
* Living related liver transplantation patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparison of patency of the bile duct between normal and Kaffes stenting. | after 6 months and after 1 year
  Comparison of patency of the bile duct 6 months after 1 year of stenting. Patency is defined as the presence of normal liver function test (direct bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (gamma-GT), alkaline phosphatase) and non-dilated bile ducts on Magnetic resonance cholangiopancreatography (MRCP). In the presence of cytomegalovirus (CMV) infection, rejection or other causes of possible disturbed liver function parameters, the MRCP findings rule over the lab tests.

SECONDARY OUTCOMES:
safety of the Kaffes stent | during a period of 1 year
  The safety of the Kaffes stent, compared to the normal stent will be assessed (e.g. change of stents, blood tests, endoscopic retrograde cholangio-pancreatography (ERCP)).
Duration of hospitalization | during a period of 1 year
Number of stent changes | during a period of 1 year
  Patients included in the plastic stenting arm will receive change of stents every 3 months for a total duration of 1 year.
  Patients included in the Kaffes stent arm will receive change of the stent every 6 months for a total duration of 1 year.
  In case the patient develops symptoms of stent occlusion (rise of liver tests, fever, septicimiae), the stent will be changed as soon as possible.
Comparison of costs between normal stenting and Kaffes stenting. | during a period of 1 year
  Comparison of costs over a period of 1 year between normal stenting and Kaffes stenting will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Van Vlierberghe, Ph.D., M.D., Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be